CLINICAL TRIAL: NCT06003218
Title: Dexmedetomidine-esketamine Combined With Oxycodone for Ultrasound-guided Percutaneous Radiofrequency Ablation in Patients With Liver Cancer: a Randomized Controlled Study
Brief Title: Dexmedetomidine-esketamine for Percutaneous Radiofrequency Liver Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023-276
Record Dates: First submitted 2023-08-12; First posted 2023-08-21 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Liver Cancer; Radiofrequency Ablation; Esketamine; Dexmedetomidine
Keywords: Liver cancer; Radiofrequency ablation; Esketamine; Dexmedetomidine
MeSH Terms: conditions — Liver Neoplasms | interventions — Remifentanil; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine-esketamine combined with oxycodone (Experimental): Dexmedetomidine-esketamine combination will be infused in addition to oxycodone; the target is to maintain a Richmond Agitation and Sedation Scale between -2 and -1 during surgery.
  Interventions: Drug: Dexmedetomidine-esketamine combination; Drug: Oxycodone
- Remifentanil combined with oxycodone (Active Comparator): Remifentanil will be infused in addition to oxycodone; the target is to maintain a Richmond Agitation and Sedation Scale between -2 and -1 during surgery.
  Interventions: Drug: Remifentanil; Drug: Oxycodone

INTERVENTIONS:
Drug: Dexmedetomidine-esketamine combination — Dexmedetomidine-esketamine mixture will be infused with doses adjusted to maintain a Richmond Agitation-Sedation Scale between -2 to -1 during surgery.
  Arms: Dexmedetomidine-esketamine combined with oxycodone
Drug: Remifentanil — Remifentanil will be infused with doses adjusted to maintain a Richmond Agitation-Sedation Scale between -2 to -1 during surgery.
  Arms: Remifentanil combined with oxycodone
Drug: Oxycodone — Oxycodone will be injected intravenously 10-15 min before puncture.

SUMMARY:
Percutaneous radiofrequency ablation is a commonly treatment for patients with liver cancer that cannot be surgically resected. During the procedure, patients need to keep awake and cooperate with the procedure, including deep breath and hold breath. However, intolerable pain generated during puncture and radiofrequency heating may cause body movements and interfere the procedure. Oxycodone is frequently used for analgesia but still insufficient. A recent study showed that dexmedetomidine-esketamine combination improves analgesia without increasing adverse events. After stopping infusion, the analgesic/sleep-promoting effects of dexmedetomidine-esketamine seemed to last for up to 24 hours.

The investigators hypothesize that dexmedetomidine-esketamine combination as a supplement to oxycodone will improve sedation and analgesia in patients undergoing radiofrequency liver ablation of the liver.

DETAILED DESCRIPTION:
Ultrasound-guided percutaneous radiofrequency ablation is a new technique to treat liver cancer. Under ultrasound guidance, a radiofrequency electrode needle is inserted into the cancer through which local high temperature is generated to coagulate and necrose the cancer tissue. Percutaneous radiofrequency ablation is currently recognized as the best treatment for patients with liver cancer that cannot be surgically resected. During the procedure, patients need to keep awake and cooperate with the procedure, including deep breath and hold breath. However, intolerable pain generated during puncture and radiofrequency heating may cause body movements and interfere the procedure.

Oxycodone is a widely used opioid. It activates the μ and κ receptors and relieves pain including visceral pain, which makes it suitable for analgesia during radiofrequency ablation. However, due to the strong stimulation of radiofrequency liver ablation, supplemental analgesics are often required to improve patient cooperation. As a commonly used supplement, remifentanil is also a μ receptor agonist that quickly reaches blood-brain balance in about 1 minute in and is rapidly hydrolyzed in tissues and blood. The problems with remifentanil are the ultra-short action and pain allergy after stopping infusion. The burning pain after percutaneous liver radiofrequency ablation may last for up to 24 hours.

Dexmedetomidine is a highly selective α2-adrenergic receptor agonist that has sedative, anxiolytic, and analgesic effects. Ketamine is a non-competitive N-methyl-D-aspartate (NMDA) receptor antagonist that is widely used in pediatric anesthesia and postoperative analgesia. Recent studies found that low-dose ketamine also has antidepressant and sleep promoting effects. Esketamine is the S-enantiomer of racemic ketamine with a higher affinity for NMDA receptors and is approximately twice as potent as racemic ketamine in analgesia. A recent study showed that dexmedetomidine-esketamine combination improves analgesia without increasing adverse events. After stopping infusion, the analgesic and sleep-promoting effects of dexmedetomidine-esketamine seemed to last for up to 24 hours.

The investigators hypothesize that dexmedetomidine-esketamine combination as a supplement to oxycodone will improve sedation and analgesia in patients undergoing radiofrequency liver ablation of the liver.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years but ≤85 years.
2. Scheduled for elective ultrasound-guided percutaneous radiofrequency ablation for primary or metastatic liver cancer.

Exclusion Criteria:

1. Refused to participate.
2. Diagnosed schizophrenia, epilepsy, Parkinson's disease, or myasthenia gravis before surgery.
3. Preoperative left ventricular ejection fraction (LVEF) <30%, or those with sick sinus syndrome, sinus bradycardia (heart rate <50 beats per minute), or atrioventricular block at grade II or above without pacemaker.
4. Diagnosed obstructive sleep apnea (OSA) or judged to be at high-risk of moderate-to-severe OSA before surgery.
5. Severe liver dysfunction (Child-Pugh grade C), severe renal dysfunction (dialysis before surgery), or classified as American Society of Anesthesiologists (ASA) grade >III before surgery.
6. Inability to communicate due to coma, severe dementia, or language barrier before surgery.
7. Allergy to any drug used during the study, or other conditions that are considered unsuitable for study participation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-09-28 (Actual)

PRIMARY OUTCOMES:
Area under curve of Numerical Rating Scale of pain during and within 24 hours after surgery. | During and within 24 hours after surgery.
  Numerical Rating Scale (NRS, an 11-point scale where 0=no pain and 10=the worst pain) of pain will be assessed after percutaneous liver puncture, start of radiofrequency-ablation, every 5±1 minutes during radiofrequency-ablation, end of radiofrequency-ablation, and 10 minutes after needle removal during surgery, as well as at 0.5, 1, 2, 3-8, >8-12h,and 24 hours after surgery.

SECONDARY OUTCOMES:
The highest Numerical Rating Scale of pain during surgery. | During surgery.
  Numerical Rating Scale (NRS, an 11-point scale where 0=no pain and 10=the worst pain) of pain will be assessed after percutaneous liver puncture, start of radiofrequency-ablation, every 2 minutes during radiofrequency-ablation, end of radiofrequency-ablation, and 10 minutes after needle removal during surgery
Number of intraoperative adjustment of study drug infusion rate. | During surgery.
  Number of adjustment of study drug infusion rate during surgery.
Number of additional oxycodone or other analgesics during and within 24 hours after surgery. | During and within 24 hours after surgery.
  Number of additional oxycodone or other analgesics during and within 24 hours after surgery.
Dose of analgesics during and within 24 hours after surgery. | During and within 24 hours after surgery.
  Dose of opioids (excluding remifentanil administered as study drugs) will be converted to intravenous morphine equivalent.
Pain intensity and opioid consumption (PIOC) index during and within 24 hours after surgery. | During and within 24 hours after surgery.
  Pain intensity will be calculated as area under curve (AUC) of Numerical Rating Scale (NRS, an 11-point scale where 0=no pain and 10=the worst pain) of pain during and within 24 hours after surgery. Opioid consumption (OC) during and within 24 hours after surgery will be calculated after excluding remifentanil administered as study drugs. Pain intensity and opioid consumption (PIOC) index will be calculated as: PIOC=[(AUCmean rank - AUCrank)/AUCmean rank] + [(OCmean rank - OCrank)/OCmean rank]. The range of the sum is -200% to +200%. Values above 0 indicate increased summed AUC and OC compared to the all patients.
Numeric Rating Scale of subjective sleep quality on the first and second nights after surgery. | On the first and second nights after surgery.
  Numerical Rating Scale (NRS, an 11-point scale where 0=the best sleep and 10=the worst sleep) of sleep quality on the first and second nights after surgery.

OTHER OUTCOMES:
Patients' evaluation on anesthesia. | Within 30 minutes after surgery.
  Patients' evaluation will be performed using the Likert five-point scale: 1=very dissatisfied, 2=dissatisfied, 3=neutral, 4=satisfied, and 5=very satisfied.
Surgeons' evaluation on anesthesia. | Within 30 minutes after surgery.
  Surgeons' evaluation will be performed using the Likert five-point scale: 1=very dissatisfied, 2=dissatisfied, 3=neutral, 4=satisfied, and 5=very satisfied.
Postoperative recovery time. | Up to 2 hours after surgery.
  Time interval between end of surgery and arrival of general ward.
Length of hospital stay after surgery. | Up to 30 days after surgery.
  Length of hospital stay after surgery.
Incidence of postoperative complications during hospital stay. | Up to 30 days after surgery.
  Postoperative complications are defined as new-onset conditions after surgery that have adverse effects on postoperative recovery and require therapeutic interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] McGahan JP, Browning PD, Brock JM, Tesluk H. Hepatic ablation using radiofrequency electrocautery. Invest Radiol. 1990 Mar;25(3):267-70. doi: 10.1097/00004424-199003000-00011. No abstract available. PMID 2185179
- [Background] European Association for Study of Liver; European Organisation for Research and Treatment of Cancer. EASL-EORTC clinical practice guidelines: management of hepatocellular carcinoma. Eur J Cancer. 2012 Mar;48(5):599-641. doi: 10.1016/j.ejca.2011.12.021. No abstract available. PMID 22424278
- [Background] Higgins H, Berger DL. RFA for liver tumors: does it really work? Oncologist. 2006 Jul-Aug;11(7):801-8. doi: 10.1634/theoncologist.11-7-801. PMID 16880239
- [Background] Olesen AE, Kristensen K, Staahl C, Kell S, Wong GY, Arendt-Nielsen L, Drewes AM. A population pharmacokinetic and pharmacodynamic study of a peripheral kappa-opioid receptor agonist CR665 and oxycodone. Clin Pharmacokinet. 2013 Feb;52(2):125-37. doi: 10.1007/s40262-012-0023-8. PMID 23212610
- [Background] Riviere PJ. Peripheral kappa-opioid agonists for visceral pain. Br J Pharmacol. 2004 Apr;141(8):1331-4. doi: 10.1038/sj.bjp.0705763. Epub 2004 Mar 29. PMID 15051626
- [Background] Wang J, Yuan X, Guo W, Xiang X, Wu Q, Fang M, Zhang W, Ding Z, Xie K, Fang J, Zhou H, Fu S. Sedation and Analgesia for Liver Cancer Percutaneous Radiofrequency Ablation: Fentanyl and Oxycodone Comparison. Int J Med Sci. 2020 Aug 12;17(14):2194-2199. doi: 10.7150/ijms.47067. eCollection 2020. PMID 32922181
- [Background] Wu WT, Jia ZY, Chen Y, Chen QF, Zu QQ, Yang ZQ, Liu S, Shi HB. The Safety and Efficacy of Oxycodone Versus Fentanyl in Percutaneous Microwave Ablation of a Liver Tumour Abutting the Capsule. Cardiovasc Intervent Radiol. 2019 Jan;42(1):87-94. doi: 10.1007/s00270-018-1980-6. Epub 2018 May 8. PMID 29740688
- [Background] Wu J, Lu Y, Cao X. Different effects of oxycodone and remifentanil in patients undergoing ultrasound-guided percutaneous radiofrequency ablation of hepatic cancer: a randomized trial. Drug Des Devel Ther. 2019 Jan 18;13:365-372. doi: 10.2147/DDDT.S188728. eCollection 2019. PMID 30705584
- [Background] Yu EH, Tran DH, Lam SW, Irwin MG. Remifentanil tolerance and hyperalgesia: short-term gain, long-term pain? Anaesthesia. 2016 Nov;71(11):1347-1362. doi: 10.1111/anae.13602. PMID 27734470
- [Background] Ongiem A, Siriussawakul A, Aungsumat Wangdee BNS W, Homsud S, Jaiyen T. Assessment of Pain Severity after Radiofrequency Ablation in Patients with Hepatocellular Carcinoma. J Med Assoc Thai. 2016 May;99(5):572-7. PMID 27501613
- [Background] Nelson LE, Lu J, Guo T, Saper CB, Franks NP, Maze M. The alpha2-adrenoceptor agonist dexmedetomidine converges on an endogenous sleep-promoting pathway to exert its sedative effects. Anesthesiology. 2003 Feb;98(2):428-36. doi: 10.1097/00000542-200302000-00024. PMID 12552203
- [Background] Xia ZQ, Chen SQ, Yao X, Xie CB, Wen SH, Liu KX. Clinical benefits of dexmedetomidine versus propofol in adult intensive care unit patients: a meta-analysis of randomized clinical trials. J Surg Res. 2013 Dec;185(2):833-43. doi: 10.1016/j.jss.2013.06.062. Epub 2013 Jul 24. PMID 23910886
- [Background] Sun YM, Zhu SN, Zhang C, Li SL, Wang DX. Effect of low-dose dexmedetomidine on sleep quality in postoperative patients with mechanical ventilation in the intensive care unit: A pilot randomized trial. Front Med (Lausanne). 2022 Aug 31;9:931084. doi: 10.3389/fmed.2022.931084. eCollection 2022. PMID 36117973
- [Background] Barrett W, Buxhoeveden M, Dhillon S. Ketamine: a versatile tool for anesthesia and analgesia. Curr Opin Anaesthesiol. 2020 Oct;33(5):633-638. doi: 10.1097/ACO.0000000000000916. PMID 32826629
- [Background] Kaur U, Pathak BK, Singh A, Chakrabarti SS. Esketamine: a glimmer of hope in treatment-resistant depression. Eur Arch Psychiatry Clin Neurosci. 2021 Apr;271(3):417-429. doi: 10.1007/s00406-019-01084-z. Epub 2019 Nov 19. PMID 31745646
- [Background] Song B, Zhu J. A Novel Application of Ketamine for Improving Perioperative Sleep Disturbances. Nat Sci Sleep. 2021 Dec 25;13:2251-2266. doi: 10.2147/NSS.S341161. eCollection 2021. PMID 34992482
- [Background] Bartova L, Papageorgiou K, Milenkovic I, Dold M, Weidenauer A, Willeit M, Winkler D, Kasper S. Rapid antidepressant effect of S-ketamine in schizophrenia. Eur Neuropsychopharmacol. 2018 Aug;28(8):980-982. doi: 10.1016/j.euroneuro.2018.05.007. Epub 2018 Jul 2. PMID 30041987
- [Background] Molero P, Ramos-Quiroga JA, Martin-Santos R, Calvo-Sanchez E, Gutierrez-Rojas L, Meana JJ. Antidepressant Efficacy and Tolerability of Ketamine and Esketamine: A Critical Review. CNS Drugs. 2018 May;32(5):411-420. doi: 10.1007/s40263-018-0519-3. PMID 29736744
- [Background] Canuso CM, Singh JB, Fedgchin M, Alphs L, Lane R, Lim P, Pinter C, Hough D, Sanacora G, Manji H, Drevets WC. Efficacy and Safety of Intranasal Esketamine for the Rapid Reduction of Symptoms of Depression and Suicidality in Patients at Imminent Risk for Suicide: Results of a Double-Blind, Randomized, Placebo-Controlled Study. Am J Psychiatry. 2018 Jul 1;175(7):620-630. doi: 10.1176/appi.ajp.2018.17060720. Epub 2018 Apr 16. PMID 29656663
- [Background] Segmiller F, Ruther T, Linhardt A, Padberg F, Berger M, Pogarell O, Moller HJ, Kohler C, Schule C. Repeated S-ketamine infusions in therapy resistant depression: a case series. J Clin Pharmacol. 2013 Sep;53(9):996-8. doi: 10.1002/jcph.122. Epub 2013 Jul 24. No abstract available. PMID 23893490
- [Background] Persson J, Hasselstrom J, Maurset A, Oye I, Svensson JO, Almqvist O, Scheinin H, Gustafsson LL, Almqvist O. Pharmacokinetics and non-analgesic effects of S- and R-ketamines in healthy volunteers with normal and reduced metabolic capacity. Eur J Clin Pharmacol. 2002 Feb;57(12):869-75. doi: 10.1007/s002280100353. PMID 11936706
- [Background] Bornemann-Cimenti H, Wejbora M, Michaeli K, Edler A, Sandner-Kiesling A. The effects of minimal-dose versus low-dose S-ketamine on opioid consumption, hyperalgesia, and postoperative delirium: a triple-blinded, randomized, active- and placebo-controlled clinical trial. Minerva Anestesiol. 2016 Oct;82(10):1069-1076. Epub 2016 Jun 21. PMID 27327855
- [Background] Hu ZC, Xu G, Zhang XW, Ma K, Jin JJ, Li PS. [Meta-analysis of the effects of dexmedetomidine combined with ketamine during dressing changes in burn patients]. Zhonghua Shao Shang Za Zhi. 2020 Jun 20;36(6):458-464. doi: 10.3760/cma.j.cn501120-20190327-00145. Chinese. PMID 32594705
- [Background] Lee KH, Lee SJ, Park JH, Kim SH, Lee H, Oh DS, Kim YH, Park YH, Kim H, Lee SE. Analgesia for spinal anesthesia positioning in elderly patients with proximal femoral fractures: Dexmedetomidine-ketamine versus dexmedetomidine-fentanyl. Medicine (Baltimore). 2020 May;99(20):e20001. doi: 10.1097/MD.0000000000020001. PMID 32443302
- [Background] Nagappa M, Wong J, Singh M, Wong DT, Chung F. An update on the various practical applications of the STOP-Bang questionnaire in anesthesia, surgery, and perioperative medicine. Curr Opin Anaesthesiol. 2017 Feb;30(1):118-125. doi: 10.1097/ACO.0000000000000426. PMID 27898430
- [Background] Andersen LPK, Gogenur I, Torup H, Rosenberg J, Werner MU. Assessment of Postoperative Analgesic Drug Efficacy: Method of Data Analysis Is Critical. Anesth Analg. 2017 Sep;125(3):1008-1013. doi: 10.1213/ANE.0000000000002007. PMID 28632527